CLINICAL TRIAL: NCT02144818
Title: GnRH Agonist Triggering Supplemented With Hcg in Women With Poor Ovarian
Brief Title: GnRH Agonist Triggering Supplemented With Hcg in Women With Poor Ovarian Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Jigal Haas MD, Senior Gynecologist and Obstetrician, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0438-JH-CTIL
Record Dates: First submitted 2014-04-28; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Women With Poor Ovarian Response
MeSH Terms: interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GnRH agonist (Active Comparator)
  Interventions: Drug: Decapeptyl
- hCG (Active Comparator)
  Interventions: Drug: Ovitrel
- dual triggering: GnRH agonist and hCG (Active Comparator)
  Interventions: Drug: Ovitrel; Drug: Decapeptyl

INTERVENTIONS:
Drug: Ovitrel — Triggering of ovulation with Ovitrel
  Arms: dual triggering: GnRH agonist and hCG; hCG
Drug: Decapeptyl — Triggering with GnRH agonist
  Arms: GnRH agonist; dual triggering: GnRH agonist and hCG

SUMMARY:
During the last decades, owing to the growing tendency of women to delay childbearing plans because of career and personal priorities, fertility specialists today are seeing more and more women with poor ovarian reserve and with poor ovarian response Controlled ovarian hyperstimulation (COH) is considered a important factor in the success of in vitro fertilization-embryo transfer (IVF-ET), enabling the recruitment of multiple oocytes and, thereby, resulting in more than one embryo. However, owing to the extreme variability in ovarian response to COH, in a subgroup of patients with poor ovarian response, this method may yield a very small number of follicles After succeeding in maximal recruitment of the follicles, the triggering of ovulation is extremely important in order to achieve, as many as, mature oocytes.

Several studies have reported retrieval of more mature oocytes after GnRH agonist triggering compared to the number of oocytes retrieved after hCG. Among the possible advantages of GnRH agonist for final oocyte maturation is the simultaneous induction of an FSH surge. The role of the natural mid-cycle FSH surge is not fully clear. FSH was reported to induce LH receptor formation in luteinizing granulosa cells, and to promote oocyte nuclear maturation and cumulus expansion .

Another method described to trigger ovulation is the "Dual triggering"- GnRH agonist 40 h prior to ovum pickup and hCG added 6 h after the first trigger. The dual triggering was described as the treatment in cases with recurrent empty follicles.

The aim of the present study is to evaluate three different methods of ovulation triggering in women with poor ovarian response

DETAILED DESCRIPTION:
Inclusion criteria:

* Women with low ovarian response according to the Bologna criteria, undergoing IVF treatments for this cause.

Exclusion criteria:

* Women with good ovarian response.
* Women with low ovarian response who are carriers of fragile X

ELIGIBILITY:
Inclusion Criteria:

* Women with low ovarian response according to the Bologna criteria, undergoing IVF treatments for this cause.

Exclusion Criteria:

* Women with good ovarian response.
* Women with low ovarian response who are carriers of fragile X

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The main outcome is the number of mature oocytes | up to 12 months
number of embryos appropriate for transfer | up to 12 month

SECONDARY OUTCOMES:
pregnancy rate | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel